CLINICAL TRIAL: NCT06146387
Title: Improved Cognitive Outcomes Associated With Feihe HMO With DHA/ARA in Infant Formula: A Randomized, Controlled Trial
Brief Title: Improved Cognitive Outcomes Associated With Feihe HMO With DHA/ARA in Infant Formula
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heilongjiang Feihe Dairy Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 22-SM-11-FEIHE-001
Record Dates: First submitted 2023-11-19; First posted 2023-11-24 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Cognitive Change
Keywords: Bayley-III Cognitive Scale; Feihe Infant Formula; HMO (Human Milk Oligosaccharides); DHA (Dehydroascorbic Acid); ARA (Arachidonic Acid)
MeSH Terms: interventions — Lactation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Two arms of participants will be assigned masked products (investigational formula and control formula) after randomization, while the participants of breastfeeding arm will not be assigned study products.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Investigational Formula (Experimental): Feihe Investigational Formula
  1. Contains 2 kinds of HMOs
  2. 5 kinds of phospholipid content reached the level of breast milk
  3. DHA&ARA reaches the content and proportion of breast milk in China
  4. Comprehensive nutrition: OPO, probiotics, lactoferrin, CPP, nucleotide, choline, inositol, taurine, L-carnitine, GOS, lutein
  Interventions: Dietary Supplement: Investigational Formula
- Control Formula (Active Comparator): Control formula contains comparable macronutrients and micronutrients, but does not contain HMO, DHA and ARA.
  Interventions: Dietary Supplement: Control Formula
- Breastfeeding (Other): breastmilk-feeding
  Interventions: Dietary Supplement: Breastfeeding

INTERVENTIONS:
Dietary Supplement: Investigational Formula — Participants in this arm will receive stage 1 and stage 2 investigational formulas. At the first (up to) 6 months, they will be fed with stage1 formula, and then switch to stage 2 formula until 12 months.
  Arms: Investigational Formula
Dietary Supplement: Control Formula — Participants in this arm will receive stage 1 and stage 2 Control formulas. At the first (up to) 6 months, they will be fed with stage1 formula, and then switch to stage 2 formula until 12 months.
  Arms: Control Formula
Dietary Supplement: Breastfeeding — Exclusively breastfed for the first 4 months and continue with supplement food without any marketed infant formula.
  Arms: Breastfeeding

SUMMARY:
The goal of this interventional clinical trial is to test the effectiveness of improving cognitive development in newly born infants fed with Feihe investigational formula product containing HMO, and DHA/ARA. The main question it aims to answer is:

- whether the score of Bayley-III cognitive scale (tested at the age of 12 months) of participants in the study product arm is significantly better than participants assigned in the other two arms.

240 qualified participants will be randomized to 3 arms (investigational formula, control formula, and breast-feeding) to consume assigned formula or breast-feeding for 12 months according to protocol. There will be up to 6 site visits arranged for each participant during the study, and all relevant clinical and questionnaire data, including the most important Barley-III cognitive scale data at the age of 12 months, will be captured, recorded and entered to CMTS (Clinical Management Trial System) for statistical analysis and reporting.

Researchers will compare the three arms to validate the assumption that the consumption of Feihe investigational formula product containing HMO, and DHA/ARA will improve cognitive development in newly born infants, along with physical development.

ELIGIBILITY:
Inclusion Criteria:

* Newborn baby, study entry before weaning (within 28 days of birth)
* Exclusively formula fed for at least 3 days prior to study entry and plan to be exclusively formula fed during the study (formula groups) OR plan to be exclusively fed with human milk during the study (breastfeeding group).
* Gestational age of 37-42 weeks (36 weeks and six days is considered 36 weeks gestational age).
* Birth weight of 2500g (5 lbs. 8 oz.) to 4200g (9 lbs. 4 oz.).
* Signed informed consent obtained for infant's participation in the study.
* Parent or guardian of the infant agrees to not enroll the infant in another interventional clinical research study while participating in this study.

Exclusion Criteria:

* History of underlying metabolic or chronic disease; congenital malformation; or any other condition which, in the opinion of the Investigator, is likely to interfere with: the ability of the infant to ingest food, the normal growth and development of the infant, or the evaluation of the infant.
* Evidence of feeding difficulties or formula intolerance, such as vomiting or poor intake, at time of randomization (at investigator discretion).
* Evidence of growth problems or concern for growth.
* Infant was born large for gestational age (LGA) (defined as birth weight-for-age exceeding 90th percentile as plotted on the growth chart provided by Feihe) from mother who was diabetic at childbirth.
* Participant is immunocompromised (according to a doctor's diagnosis of immunodeficiency such as Combined Immunodeficiencies, DiGeorge Syndrome, Wiskott-Aldrich Syndrome, Severe Congenital Neutropenia and Secondary Immunodeficiencies linked to HIV infection, Down Syndrome or others) and children with known head/brain disease/injury.
* Use of probiotics/prebiotics before the study.

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 240 (Actual)
Dates: Start 2023-11-14 (Actual); Primary Completion 2025-04-03 (Actual); Study Completion 2025-04-03 (Actual)

PRIMARY OUTCOMES:
Bayley-III cognitive scale | At the age of 12 months
  Cognitive Scale of the Bayley Scales of Infant and Toddler Development, Third Edition (BSID-III) is used to evaluate the cognitive development level of participants at the age of 12 months.
  Bayley-III contains two scoring systems of composite scores and percentile ranks. The normal range for composite scores is between 40-160 with mean at 100 and 0-99 for the percentile ranks.
  Higher scores mean a better outcome.

SECONDARY OUTCOMES:
Weight in grams | At the age of 15-28 days and 3, 6, 9, 12 months
  The weight measurement (gram) of the participant for each site visit
Height in cm | At the age of 15-28 days and 3, 6, 9, 12 months
  The height measurement (cm) of the participant for each site visit
Head circumference in cm | At the age of 15-28 days and 3, 6, 9, 12 months
  The head circumference measurement (cm) of the participant for each site visit
Amount of formula intake in ml | At the age of 15-28 days and 3, 6, 9, 12 months
  The 24-Hour dietary recall of Formula intake (amount in ml of study formula, any other infant formula or milk consumed) of the participant for each site visit
Stool Characteristics Questionnaire | At the age of 15-28 days and 3, 6 months
  The frequency of bowel movements and the rating score (0-5) of the stool consistency over the 24-hour period. The rating score of the stool consistency from the stool picture:
  (0) No bowel movement;
  1. Hard- dry, hard pellets;
  2. Formed- definite shape, not dry;
  3. Soft-no definite shape, pasty;
  4. Unformed or seedy- no shape, some water or small lumps ;
  5. Waterly- no shape, mainly water
  where the score of 0-1 represents poor stool characteristics, while 2-5 represents fine stool characteristics.
Medically-confirmed adverse events | baseline day to 12 months
  The frequency of medically-confirmed adverse events occurred during the study

CONTACTS AND LOCATIONS:
Overall Officials: Yajun Xu, MD, Principal Investigator — Peking University
Locations (3):
- China (3):
  - Jinhua Nanyuan Community Health Center (site 1919), Jinhua, Zhejiang
  - Li Pu Community Hospital, Jinhua, Zhejiang
  - Qiu Bin Community Hospital, Jinhua, Zhejiang